CLINICAL TRIAL: NCT04950959
Title: Observational Post-Market Study of the XACT ACE Robotic System
Brief Title: XACT ACE Observational Registry
Status: Recruiting | Type: Observational
Sponsor: Xact Robotics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-REG-01-2020
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Tumors
Keywords: CT-guided percutaneous procedure; Percutaneous biopsy; XACT ACE Robotic System
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: Subjects undergoing CT-guided, minimally invasive percutaneous procedures in an interventional radiology setting
  Interventions: Device: Hands-free, user-controlled robotic system intended to assist in the planning and advancement of an instrument during CT guided percutaneous procedures. T

INTERVENTIONS:
Device: Hands-free, user-controlled robotic system intended to assist in the planning and advancement of an instrument during CT guided percutaneous procedures. T — The system is used for trajectory planning and is intended to assist the physician in the positioning of an instrument, such as a needle, where CT imaging is used for target trajectory planning and intraoperative tracking. The XACT ACE Robotic System uses a computerized quantitative guidance system, which provides real-time, accurate needle guidance, including advancement and steering of the needle from the entry point on the subject's body to the target point within the body.

SUMMARY:
Compile real world data on the use of the XACT ACE Robotic System

DETAILED DESCRIPTION:
The purpose of this observational post-market study is to compile real world data on the use of the XACT ACE Robotic System in subjects undergoing CT guided, minimally invasive percutaneous procedures.

The objectives are to 1) evaluate the proportion of procedures in which the instrument reached the pre-defined target, based on the physician's determination and CT imaging confirmation, 2) To evaluate system accuracy defined as the measured distance from the tip of the instrument to the target location at the at the end of the instrument insertion, and 3) Incidence of intra- and post-procedural adverse events.

Up to 500 patients will be enrolled in this multicenter, nonrandomized, single arm registry.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Subjects undergoing CT-guided, minimally invasive percutaneous procedures in the interventional radiology suite
3. Subject is willing to sign informed consent for the purposes of data collection

Exclusion Criteria:

1. No exclusion criteria other than listed in the product Instructions for Use (IFU)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing CT guided, minimally invasive percutaneous procedures in an interventional radiology setting.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of successful procedures | 1 hour
  To evaluate the proportion of procedures in which the instrument reached the pre-defined target based on the physician's determination and CT imaging confirmation.
System accuracy | 1 hour
  To evaluate system accuracy defined as the measured distance from the tip of the instrument to the target location at the end of the instrument insertion.
Assessment of Safety | 2 hours post-procedure
  Incidence of intra- and post-procedural events

CONTACTS AND LOCATIONS:
Overall Officials: Mark Macedo, Study Director — XACT Robotics
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No